CLINICAL TRIAL: NCT02295813
Title: A Single Center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Pharmacokinetics of One Single Intravenous Dose and 5-day Repeated Intravenous Doses of FBF001 in Healthy Male Subjects
Brief Title: Safety and Pharmacokinetics Study of FBF001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fab'entech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201101H-TOLPKE
Record Dates: First submitted 2014-11-12; First posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Avian Influenza
MeSH Terms: conditions — Influenza in Birds | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- FBF001 (Experimental): FBF001 must be administered by intravenous route during 1 hour. The dose must be calculated according to the body weight of the subject and diluted in sodium chloride 0.9%.
  FBF001 is administered once during 1 day or once per day during 5 days.
  Interventions: Biological: FBF001
- Placebo (Placebo Comparator): The placebo must be administered by intravenous route during 1 hour. It administered once during 1 day or once per day during 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: FBF001
  Arms: FBF001
Drug: Placebo
  Other Names: Sodium chloride 0.9%
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the clinical and laboratory safety and to determine the pharmacokinetic profile of FBF001.

ELIGIBILITY:
Inclusion Criteria:

* subject between 21-40 years old
* with body mass index in the range 18 to 30 Kg/m2

Exclusion Criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, haematological, neurological, osteo-muscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness
* Any vaccination within three months before the inclusion
* Any vaccination against H5N1 virus
* Planned receipt of any vaccine during the study
* Any infectious disease within the month before the inclusion
* Any history of animal proteins allergy, animal allergy and/or any drug, food and pollen allergy
* Who has received blood or plasma derivatives (human or animal) in the three months preceding the initiation of the study
* Any medication within 14 days before the inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of that drug

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure | The subjects will be followed during their hospitalization stay (2 days or 6 days) and up to an average of 3 weeks after hospitalization
  mmHg
ECG evaluation | The subjects will be followed during their hospitalization stay (2 days or 6 days) and up to an average of 3 weeks after hospitalization
  12-lead ECG
Haematology | The subjects will be followed during their hospitalization stay (2 days or 6 days) and up to an average of 3 weeks after hospitalization
  Normal values of haematology parameters
Complement activation assay | Before dosing, at the end of infusion and 2hours after the beginning
  ng/mL
Heart rate | The subjects will be followed during their hospitalization stay (2 days or 6 days) and up to an average of 3 weeks after hospitalization
  bpm
Oral temperature | The subjects will be followed during their hospitalization stay (2 days or 6 days) and up to an average of 3 weeks after hospitalization
  Celcius degree
Body weight | The subjects will be followed during their hospitalization stay (2 days or 6 days) and up to an average of 3 weeks after hospitalization
  kg
Blood chemistry | The subjects will be followed during their hospitalization stay (2 days or 6 days) and up to an average of 3 weeks after hospitalization
  Normal values of blood chemistry parameters

REFERENCES:
- [Derived] Bal C, Herbreteau CH, Buchy P, Rith S, Zaid M, Kristanto W, Han V, Reynaud C, Granjard P, Lepine B, Durand C, Tambyah PA. Safety, potential efficacy, and pharmacokinetics of specific polyclonal immunoglobulin F(ab')(2) fragments against avian influenza A (H5N1) in healthy volunteers: a single-centre, randomised, double-blind, placebo-controlled, phase 1 study. Lancet Infect Dis. 2015 Mar;15(3):285-92. doi: 10.1016/S1473-3099(14)71072-2. Epub 2015 Feb 5. PMID 25662592